CLINICAL TRIAL: NCT00698737
Title: Reducing Cocaine/Heroin Abuse With SR-Amphetamine and Buprenorphine (ARC)
Brief Title: Treatment Study: Reducing Cocaine/Heroin Abuse With SR-Amphetamine and Buprenorphine (ARC)
Acronym: ARC
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Principal Investigator, Wayne State University
Other Study IDs: NIDA 022243-2; R01DA022243 (NIH); DPMCDA (Other: NIDA)
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Heroin Dependence; Opioid-Related Disorders; Cocaine Abuse or Dependence
Keywords: Opioid; Cocaine
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders; Cocaine-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This research study takes place at Wayne State University and will take about 11 weeks to complete. This is a treatment research study for individuals who currently have cocaine abuse or dependence, and who may also have heroin dependence. The purpose of this study is to test whether oral sustained release d-amphetamine (SR-AMP) is safe and more effective than placebo for preventing relapse to cocaine use for individuals who abuse or are dependent upon cocaine. We are also interested whether, for patients who are dependent on cocaine and heroin, whether SR-AMP is safe and effective for preventing cocaine relapse in combination with buprenorphine.

DETAILED DESCRIPTION:
Cocaine dependence, particularly in combination with heroin dependence, poses serious and substantial public health, social, and economic problems (e.g., high medical costs, crime, lost productivity). Cocaine and heroin use disorders often co-occur, and this conjunction is associated with higher rates of medical and psychiatric problems and worse drug abuse treatment outcome.

Many medications have been tested, but have failed, for treating cocaine dependence alone or in cocaine abusers who also use heroin.

This clinical trial will test whether SR-AMP is more effective than placebo for preventing relapse to cocaine use, using SR-AMP for patients with only cocaine dependence, or in combination with buprenorphine (for those patients who are also dependent on heroin).

Participants will first be an outpatient and must come to the Jefferson Avenue Research Program three times per week (e.g. Monday, Wednesday, Friday) to measure drug use and drug-related symptoms. This phase will last at least 2 weeks.

Next, participants will live on an inpatient research unit for seven (7) consecutive nights. During the weeklong inpatient stay, in addition to receiving SR-AMP or placebo capsules, participants will begin counseling treatment to help prepare to avoid relapse after they are discharged from the inpatient unit.

After the inpatient stay, participants will then be an outpatient and come to the Jefferson Ave. Research Program daily for eight (8) weeks. Throughout all eight weeks, three urine samples will be collected each week to assess illicit drug use, and questionnaires related to drug symptoms and to assess mood and risk behaviors will be given.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant and non-lactating females between 18-55 years of age who are seeking treatment for their drug use.
* Females of childbearing potential are eligible to participate if using an acceptable method of birth control.
* All participants must be free from any significant clinical abnormalities based on medical history, physical examination, ECG, and screening laboratory tests.
* Participants must weigh at least 50kg (110lbs).
* Participants must meet DSM-IV criteria for current Cocaine Abuse or Dependence, and possibly Opioid Dependence, and provide a cocaine positive (and, if opioid dependent, opioid positive) urine sample.
* Participants will not be excluded if they meet DSM-IV criteria for current Alcohol or Sedative Abuse (but they will be excluded for current Alcohol or Sedative Dependence).
* Participants must not be under the influence of alcohol (BAL <.002) and sign informed consent during screening.

Exclusion Criteria:

* Volunteers will not be eligible for this study if they present with psychiatric illness, neurological disease, cardiovascular disease, pulmonary disease, systemic disease, other current substance dependence (except cocaine, heroin or nicotine).
* If they are cognitively impaired, currently being treated for Cocaine or Opioid Dependence, using prohibited medications, or females who are pregnant, lactating, or if heterosexually active not using medically approved birth control measures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Heroin dependent and Cocaine abuse or dependent research volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2008-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Derived] Stoltman JJ, Woodcock EA, Lister JJ, Greenwald MK, Lundahl LH. Exploration of the telescoping effect among not-in-treatment, intensive heroin-using research volunteers. Drug Alcohol Depend. 2015 Mar 1;148:217-20. doi: 10.1016/j.drugalcdep.2015.01.010. Epub 2015 Jan 19. PMID 25630964